CLINICAL TRIAL: NCT01806883
Title: Evaluation of the Effects of Rehabilitation Using the "Wii" on Upper Limb Kinematics in Chronic Stroke Patients.
Acronym: WII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P110701
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Post-stroke Hemiparetic Patients (at Least 6 Months Post Stroke); Age Between 18-75 Years
Keywords: Hemiparesis,; Rehabilitation,; WII,; Upper limb,; Movement strategies.
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation using Nintendo-Wii (Experimental): 30 patients will receive rehabilitation using Nintendo-Wii.
  Interventions: Behavioral: WII Rehabilitation
- Traditional physiotherapy (Active Comparator): 30 patients will receive traditional physiotherapy.
  Interventions: Behavioral: Traditional rehabilitation

INTERVENTIONS:
Behavioral: WII Rehabilitation — 30 patients will receive "Wii" rehabilitation of 15 minutes (tennis, boxing and golf), in comparison with 10 healthy subjects.
  Arms: Rehabilitation using Nintendo-Wii
Behavioral: Traditional rehabilitation — 30 patients will receive the traditional rehabilitation.
  Arms: Traditional physiotherapy

SUMMARY:
The purpose of this study is to evaluate changes in strategies of hemiparetic upper limb movement in chronic stroke patients following rehabilitation using the "Nintendo Wii". The investigators hypothesize that patients will increase their use of compensatory strategies following this rehabilitation.

DETAILED DESCRIPTION:
The principal aim of this study is to evaluate changes in strategies of hemiparetic upper limb movement in chronic stroke patients following twelve one hour sessions of rehabilitation using the "Nintendo Wii" over a period of four weeks, and to compare with a group of patients receiving traditional upper limb rehabilitation of the same duration. The investigators hypothesize that the use of compensatory strategies will increase in the group receiving the "Wii" rehabilitation while they will decrease in the group receiving traditional rehabilitation. The investigators further hypothesize that this will have an impact on the functional benefit with a greater improvement of function in the group receiving traditional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 75 years Right handed Hemiparesis following vascular lesions of a single hemisphere of more than 6 months duration.

Not a regular 'Wii' user Able to bring the hand to the mouth. No botulinum toxin injections within the previous 3 months Having given informed consent

Exclusion Criteria:

Major cognitive or perceptive deficits Cerebellar syndrome Epileptic fits within the previous year Pacemaker user Un-corrected visual deficits No social security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Degree of elbow extension during an active reaching task | 6 minutes

SECONDARY OUTCOMES:
Clinical | 1 hour and half
  Pain (VAS) (evaluated at the beginning and end of each session) Borg scale of perceived effort (evaluated at the end of each session) Fugl-Meyer (upper limb section) (evaluated before and after the rehabilitation period) Box and Block test (evaluated before and after the rehabilitation period) Action Research Arm Test (ARAT) (evaluated before and after the rehabilitation period) Motor Activity Log (MAL) (evaluated before and after the rehabilitation period) Stroke Impact scale (SIS) (evaluated before and after the rehabilitation period) Satisfaction (VAS) (evaluated at the end of the rehabilitation period)
Kinematic measures | 45 minutes
  Parameters relating to hand trajectory (smoothness, curvature, velocity) and upper limb joint angles (trunk flexion, shoulder abduction) during an active reaching task using an electromagnetic motion capture system. (evaluated before and after the rehabilitation period)
Kinetic measures | 45 minutes
  Capacity to regulate grip force during a visuo-motor task using an instrumented device. (evaluated before and after the rehabilitation period)
Movement strategies during 'Wii rehabilitation' | 45 minutes
  The number and extent of the movements made with the upper limb during 'wii rehabilitation' will be recorded using accelerometers.
MRI | 1 hour
  The extent and localization of the lesions will be evaluated using MRIcro and correlations will be sought between the lesion locations and the kinematic and kinetic characteristics of the patients.
  Evaluations will be carried out during the week preceding and the week following the rehabilitation period. The evaluating therapist will be blinded to the type of rehabilitation received by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Djamel Bensmail, MD, Principal Investigator — Physical medicine and rehabilation Department, Hôpital RAYMOND POINCARE, 92380 Garches, France
Locations (1):
- Djamel Bensmail, Garches, Hauts-de-Seine, France

REFERENCES:
- [Derived] Teremetz M, Garcia Alvarez A, Hanneton S, Roby-Brami A, Roche N, Bensmail D, Lindberg P, Robertson JVG. Improving upper-limb and trunk kinematics by interactive gaming in individuals with chronic stroke: A single-blinded RCT. Ann Phys Rehabil Med. 2022 May;65(3):101622. doi: 10.1016/j.rehab.2021.101622. Epub 2022 Feb 26. PMID 34929355